CLINICAL TRIAL: NCT02615860
Title: Efficacy and Safety of Topical Trichloroacetic Acid vs. Electrocautery for the Treatment of Anal Intraepithelial Neoplasia in HIV-positive Patients (TECAIN) - a Randomized Controlled Trial
Brief Title: Efficacy and Safety of TCA vs. ECA for the Treatment of AIN in HIV-positive Patients
Acronym: TECAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Stefan Esser M.D., Dr. med., University Hospital, Essen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01KG1425
Record Dates: First submitted 2015-11-19; First posted 2015-11-26 (Estimated); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Anal Intraepithelial Neoplasia (AIN) in HIV-infected Patients
Keywords: HIV-infection; anal cancer (AC); anal cancer prevention; anal dysplasia; anal intraepithelial neoplasia (AIN); human papillomavirus (HPV); HPV-induced anal cancer precursor lesions; electrocautery (ECA); topical trichloroacetic acid (TCA) treatment.
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Anus Neoplasms | interventions — Trichloroacetic Acid; Therapeutics; Electrocoagulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Topical 85% trichloroacetic acid (TCA) (Experimental): AIN lesions are treated with trichloric acid
  Interventions: Other: Topical 85% trichloroacetic acid (TCA)
- Surgical electrocautery (ECA) (Active Comparator): AIN lesions are treated with electrocautery
  Interventions: Procedure: Surgical electrocautery (ECA)

INTERVENTIONS:
Other: Topical 85% trichloroacetic acid (TCA) — In the experimental intervention arm, all visible lesions are treated with 85% TCA by dipping the wooden stick end of a cotton swab into a cup containing TCA. The stick end is saturated with TCA and is inserted through the anoscope and directed to the lesion under HRA guidance. TCA is applied to the lesion repeatedly until the lesion changes to a dense white colour. Each TCA application session is followed by another appointment four weeks later, where the clinician re-evaluates the lesions of the patient and determines whether a next TCA application is necessary up to a maximum of four times
  Other Names: Topical treatment with trichloroacetic acid (TCA)
  Arms: Topical 85% trichloroacetic acid (TCA)
Procedure: Surgical electrocautery (ECA) — In the control arm, HRA-guided ECA, is performed every 4 weeks up to a maximum of four times. All visible lesions are ablated at every visit. Bleeding from small vessels can be stopped by ECA. Patients undergo local anaesthesia if necessary
  Other Names: Device: Electrocauter
  Arms: Surgical electrocautery (ECA)

SUMMARY:
Comparative evaluation of efficacy and safety of high-resolution anoscopy (HRA)-guided topical treatment (trichloroacetic acid, TCA) vs. surgical treatment (electrocautery, ECA) in HIV-positive patients for human papillomavirus (HPV)- induced AIN, an anal cancer precursor. The primary hypothesis is that cost-saving and simple TCA treatment is non-inferior to the current best option therapy with ECA. TCA treatment would also be possible in the normal setting of a doctor´s office without extensive specialization and without complex technical equipment.

DETAILED DESCRIPTION:
Anal human papillomavirus (HPV)-infection and HPV-induced AIN, an anal cancer precursor, are very frequent in HIV-positive patients (HIV+), especially in men who have sex with men (MSM), but also in women. Consequently, HIV+ have a strongly increased risk for anal cancer. Screening for and treatment of AIN are recommended in HIV+, although only two RCT on AIN treatment have been published. We plan a multicenter, unblinded, non-inferiority RCT that evaluates the efficacy and safety of 2 high-resolution anoscopy (HRA)-guided treatment options for AIN: topical application of trichloroacetic acid (TCA) and surgical treatment with electrocautery (ECA).

ECA was the best option for intra-anal AIN in a recent randomized controlled trial (RCT). TCA, an inexpensive and established therapy for genital warts, has been evaluated for AIN only in a retrospective pilot study that showed clearance rates comparable to those found for ECA, with possibly less adverse events (AE). Our primary hypothesis is that cost-saving and simple TCA is non-inferior to ECA. 2800 HIV+ will be screened by HRA in 9 proctological centers and 560 HIV+ with histologically confirmed intra-anal AIN will be randomized (1:1) to receive up to 4 treatments with TCA or ECA within 12 weeks. The primary efficacy endpoint is clinical (HRA) and histological resolution of AIN 4 weeks after the last treatment. Secondary endpoints comprise recurrence of AIN 24 weeks after end of therapy, the number of interventions, AE, and the influence of HPV parameters such as anal HPV-types, viral load and HPV-oncogene-mRNA.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive patients
* Legally eligible patients and age ≥ 18 years
* Sufficient knowledge of the German language, spoken and written
* Patient is willing and able to appear regularly to the treatment- and follow-up appointments
* Clinically visible AIN-lesion, which was confirmed by histopathology (findings not older than 2 weeks after the date of collection and removal date no longer than 16 weeks prior to baseline)
* Written informed consent

Exclusion Criteria:

* Currently diagnosed anal cancer or anal cancer in anamnesis (within the last 5 years)
* Acute life-threatening disease
* Participation in a proctologic study within the last 30 days
* Participation in this study at an earlier date
* Simultaneous participation in another clinical trial, which excludes the participation in this study
* Simultaneous topical and systemic treatments wtih medications that affect the study outcome, such as immunomodulatory substances: Interferone, imiquimod or systemic glucocorticosteroids
* lactation
* Pregnancy: In patients of childbearing age, a pregnancy has to be ruled out by pregnancy test or other suitable methods.
* Women of childbearing potential without adequate contraceptive protection.
* Contraindication for using trichloroacetic acid or electrocautery
* Patients in whom general anesthesia in the treatment of AIN is necessary already at study start
* Other serious intra-anal and proctologic disorders, which make additional proctologic or systemic treatments necessary, which influence the study result, such as an active Crohn's disease, which must be treated locally and systemically with immunosuppressives or an active proctitis.
* Patients who have been vaccinated before baseline against HPV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Therapeutic success (success rate) defined as clinically (HRA) and histologically confirmed resolution (normal histology) or regression (from AIN2/3 to AIN1) of AIN | Four weeks after the last treatment within TECAIN
  The primary endpoint is therapeutic success (success rate) defined as clinically (HRA) and histologically confirmed resolution (normal histology) or regression (from AIN 2/3 to AIN1) of AIN four weeks after the last treatment within TECAIN. Patients not showing up at this mandatory follow-up appointment will be counted as treatment failure. Histologically confirmed resolution/regression 4 (to 8) weeks after therapy has been the primary endpoint in the two published RCTs and in several pilot studies. Clearance of AIN after treatment is the most relevant endpoint for patients, since AIN can rapidly progress to AC in HIV+ patients.

SECONDARY OUTCOMES:
Recurrence of AIN at the previously treated sites | 24 weeks after the end of TECAIN treatment
Number of interventions needed during the 12 weeks TECAIN treatment period. | 4 weeks after the end of TECAIN treatment
  Additional treatments are possible after baseline, but they are not mandatory, if the lesions are cleared. So 4 weeks after each treatment the investigator checks, if the lesions are cleared and decides if he does another treatment or if the patient can progress to the follow up
Pain of the proctologic AIN treatments | Up to 16 weeks after study start
  Additional treatments are possible after baseline, but they are not mandatory, if the lesions are cleared. So 4 weeks after each treatment the investigator checks, if the lesions are cleared and decides if he does another treatment or if the patient can progress to the follow up
Anal HPV types, HPV multiplicity, HPV DNA load and HPV oncogene mRNA | Baseline, 4 and 24 weeks after the end of TECAIN treatment
Recurrence of AIN or new lesions | 6 months after completion of TECAIN treatment in previously treated areas
Duration of treatment phase | 24 weeks after the end of TECAIN treatment
Adverse events | During the whole study up to 36 weeks
Treatment costs | 24 weeks after the end of TECAIN treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinikum Essen, Klinik für Dermatologie, Essen, Nordrheinwestfalen, Germany

REFERENCES:
- [Background] Berry JM, Jay N, Cranston RD, Darragh TM, Holly EA, Welton ML, Palefsky JM. Progression of anal high-grade squamous intraepithelial lesions to invasive anal cancer among HIV-infected men who have sex with men. Int J Cancer. 2014 Mar 1;134(5):1147-55. doi: 10.1002/ijc.28431. Epub 2013 Sep 14. PMID 23934991
- [Background] de Pokomandy A, Rouleau D, Ghattas G, Trottier H, Vezina S, Cote P, Macleod J, Allaire G, Hadjeres R, Franco EL, Coutlee F. HAART and progression to high-grade anal intraepithelial neoplasia in men who have sex with men and are infected with HIV. Clin Infect Dis. 2011 May;52(9):1174-81. doi: 10.1093/cid/cir064. Epub 2011 Mar 1. PMID 21364075
- [Background] Fox PA, Nathan M, Francis N, Singh N, Weir J, Dixon G, Barton SE, Bower M. A double-blind, randomized controlled trial of the use of imiquimod cream for the treatment of anal canal high-grade anal intraepithelial neoplasia in HIV-positive MSM on HAART, with long-term follow-up data including the use of open-label imiquimod. AIDS. 2010 Sep 24;24(15):2331-5. doi: 10.1097/QAD.0b013e32833d466c. PMID 20729710
- [Background] Fox PA. Treatment options for anal intraepithelial neoplasia and evidence for their effectiveness. Sex Health. 2012 Dec;9(6):587-92. doi: 10.1071/SH11157. PMID 22951292
- [Background] Goldie SJ, Kuntz KM, Weinstein MC, Freedberg KA, Welton ML, Palefsky JM. The clinical effectiveness and cost-effectiveness of screening for anal squamous intraepithelial lesions in homosexual and bisexual HIV-positive men. JAMA. 1999 May 19;281(19):1822-9. doi: 10.1001/jama.281.19.1822. PMID 10340370
- [Background] Heitland W, Schadlich PK, Chen X, Remy V, Moro L. Annual cost of hospitalization, inpatient rehabilitation and sick leave of anal cancer in Germany. J Med Econ. 2013;16(3):364-71. doi: 10.3111/13696998.2012.759582. Epub 2013 Jan 2. PMID 23253056
- [Background] Hessol NA, Holly EA, Efird JT, Minkoff H, Weber KM, Darragh TM, Burk RD, Strickler HD, Greenblatt RM, Palefsky JM. Concomitant anal and cervical human papillomavirusV infections and intraepithelial neoplasia in HIV-infected and uninfected women. AIDS. 2013 Jul 17;27(11):1743-51. doi: 10.1097/QAD.0b013e3283601b09. PMID 23803793
- [Background] Julious SA, Campbell MJ. Tutorial in biostatistics: sample sizes for parallel group clinical trials with binary data. Stat Med. 2012 Oct 30;31(24):2904-36. doi: 10.1002/sim.5381. Epub 2012 Jun 19. PMID 22714646
- [Background] Kreuter A, Potthoff A, Brockmeyer NH, Gambichler T, Stucker M, Altmeyer P, Swoboda J, Pfister H, Wieland U; German Competence Network HIV/AIDS. Imiquimod leads to a decrease of human papillomavirus DNA and to a sustained clearance of anal intraepithelial neoplasia in HIV-infected men. J Invest Dermatol. 2008 Aug;128(8):2078-83. doi: 10.1038/jid.2008.24. Epub 2008 Feb 14. PMID 18273049
- [Background] Kreuter A, Wieland U. Human papillomavirus-associated diseases in HIV-infected men who have sex with men. Curr Opin Infect Dis. 2009 Apr;22(2):109-14. doi: 10.1097/QCO.0b013e3283229fc8. PMID 19276878
- [Background] Kreuter A, Potthoff A, Brockmeyer NH, Gambichler T, Swoboda J, Stucker M, Schmitt M, Pfister H, Wieland U; German Competence Network HIV/AIDS. Anal carcinoma in human immunodeficiency virus-positive men: results of a prospective study from Germany. Br J Dermatol. 2010 Jun;162(6):1269-77. doi: 10.1111/j.1365-2133.2010.09712.x. Epub 2010 Feb 22. PMID 20184584
- [Background] Lam JM, Hoch JS, Tinmouth J, Sano M, Raboud J, Salit IE. Cost-effectiveness of screening for anal precancers in HIV-positive men. AIDS. 2011 Mar 13;25(5):635-42. doi: 10.1097/QAD.0b013e3283434594. PMID 21139488
- [Background] Legarth R, Helleberg M, Kronborg G, Larsen CS, Pedersen G, Pedersen C, Jensen J, Nielsen LN, Gerstoft J, Obel N. Anal carcinoma in HIV-infected patients in the period 1995-2009: a Danish nationwide cohort study. Scand J Infect Dis. 2013 Jun;45(6):453-9. doi: 10.3109/00365548.2012.737476. Epub 2013 Jan 7. PMID 23294033
- [Background] Macaya A, Munoz-Santos C, Balaguer A, Barbera MJ. Interventions for anal canal intraepithelial neoplasia. Cochrane Database Syst Rev. 2012 Dec 12;12(12):CD009244. doi: 10.1002/14651858.CD009244.pub2. PMID 23235673
- [Background] Machalek DA, Poynten M, Jin F, Fairley CK, Farnsworth A, Garland SM, Hillman RJ, Petoumenos K, Roberts J, Tabrizi SN, Templeton DJ, Grulich AE. Anal human papillomavirus infection and associated neoplastic lesions in men who have sex with men: a systematic review and meta-analysis. Lancet Oncol. 2012 May;13(5):487-500. doi: 10.1016/S1470-2045(12)70080-3. Epub 2012 Mar 23. PMID 22445259
- [Background] Orchard M, Roman A, Parvaiz AC. Anal intraepithelial neoplasia--is treatment better than observation? Int J Surg. 2013;11(6):438-41. doi: 10.1016/j.ijsu.2013.04.011. Epub 2013 May 2. PMID 23643642
- [Background] Palefsky JM, Holly EA, Efirdc JT, Da Costa M, Jay N, Berry JM, Darragh TM. Anal intraepithelial neoplasia in the highly active antiretroviral therapy era among HIV-positive men who have sex with men. AIDS. 2005 Sep 2;19(13):1407-14. doi: 10.1097/01.aids.0000181012.62385.4a. PMID 16103772
- [Background] Palefsky JM. Anal cancer prevention in HIV-positive men and women. Curr Opin Oncol. 2009 Sep;21(5):433-8. doi: 10.1097/CCO.0b013e32832f511a. PMID 19587592
- [Background] Piketty C, Selinger-Leneman H, Bouvier AM, Belot A, Mary-Krause M, Duvivier C, Bonmarchand M, Abramowitz L, Costagliola D, Grabar S. Incidence of HIV-related anal cancer remains increased despite long-term combined antiretroviral treatment: results from the french hospital database on HIV. J Clin Oncol. 2012 Dec 10;30(35):4360-6. doi: 10.1200/JCO.2012.44.5486. Epub 2012 Oct 22. PMID 23091098
- [Background] Richel O, Wieland U, de Vries HJ, Brockmeyer NH, van Noesel C, Potthoff A, Prins JM, Kreuter A. Topical 5-fluorouracil treatment of anal intraepithelial neoplasia in human immunodeficiency virus-positive men. Br J Dermatol. 2010 Dec;163(6):1301-7. doi: 10.1111/j.1365-2133.2010.09982.x. Epub 2010 Nov 4. PMID 20716208
- [Background] Richel O, de Vries HJ, van Noesel CJ, Dijkgraaf MG, Prins JM. Comparison of imiquimod, topical fluorouracil, and electrocautery for the treatment of anal intraepithelial neoplasia in HIV-positive men who have sex with men: an open-label, randomised controlled trial. Lancet Oncol. 2013 Apr;14(4):346-53. doi: 10.1016/S1470-2045(13)70067-6. Epub 2013 Mar 15. PMID 23499546
- [Background] Sanclemente G, Herrera S, Tyring SK, Rady PL, Zuleta JJ, Correa LA, He Q, Wolff JC. Human papillomavirus (HPV) viral load and HPV type in the clinical outcome of HIV-positive patients treated with imiquimod for anogenital warts and anal intraepithelial neoplasia. J Eur Acad Dermatol Venereol. 2007 Sep;21(8):1054-60. doi: 10.1111/j.1468-3083.2007.02169.x. PMID 17714124
- [Background] Silling S, Kreuter A, Hellmich M, Swoboda J, Pfister H, Wieland U. Human papillomavirus oncogene mRNA testing for the detection of anal dysplasia in HIV-positive men who have sex with men. J Clin Virol. 2012 Apr;53(4):325-31. doi: 10.1016/j.jcv.2011.12.029. Epub 2012 Jan 18. PMID 22261122
- [Background] Silverberg MJ, Lau B, Justice AC, Engels E, Gill MJ, Goedert JJ, Kirk GD, D'Souza G, Bosch RJ, Brooks JT, Napravnik S, Hessol NA, Jacobson LP, Kitahata MM, Klein MB, Moore RD, Rodriguez B, Rourke SB, Saag MS, Sterling TR, Gebo KA, Press N, Martin JN, Dubrow R; North American AIDS Cohort Collaboration on Research and Design (NA-ACCORD) of IeDEA. Risk of anal cancer in HIV-infected and HIV-uninfected individuals in North America. Clin Infect Dis. 2012 Apr;54(7):1026-34. doi: 10.1093/cid/cir1012. Epub 2012 Jan 30. PMID 22291097
- [Background] Singh JC, Kuohung V, Palefsky JM. Efficacy of trichloroacetic acid in the treatment of anal intraepithelial neoplasia in HIV-positive and HIV-negative men who have sex with men. J Acquir Immune Defic Syndr. 2009 Dec 1;52(4):474-9. doi: 10.1097/QAI.0b013e3181bc0f10. PMID 19779306
- [Background] Solomon D, Davey D, Kurman R, Moriarty A, O'Connor D, Prey M, Raab S, Sherman M, Wilbur D, Wright T Jr, Young N; Forum Group Members; Bethesda 2001 Workshop. The 2001 Bethesda System: terminology for reporting results of cervical cytology. JAMA. 2002 Apr 24;287(16):2114-9. doi: 10.1001/jama.287.16.2114. PMID 11966386
- [Background] Steele SR, Varma MG, Melton GB, Ross HM, Rafferty JF, Buie WD; Standards Practice Task Force of the American Society of Colon and Rectal Surgeons. Practice parameters for anal squamous neoplasms. Dis Colon Rectum. 2012 Jul;55(7):735-49. doi: 10.1097/DCR.0b013e318255815e. No abstract available. PMID 22706125
- [Background] van der Zee RP, Richel O, de Vries HJ, Prins JM. The increasing incidence of anal cancer: can it be explained by trends in risk groups? Neth J Med. 2013 Oct;71(8):401-11. PMID 24127500
- [Background] Vogel M, Friedrich O, Luchters G, Holleczek B, Wasmuth JC, Anadol E, Schwarze-Zander C, Nattermann J, Oldenburg J, Sauerbruch T, Rockstroh JK, Spengler U. Cancer risk in HIV-infected individuals on HAART is largely attributed to oncogenic infections and state of immunocompetence. Eur J Med Res. 2011 Mar 28;16(3):101-7. doi: 10.1186/2047-783x-16-3-101. PMID 21486722
- [Background] Wieland U, Kreuter A. One step towards standardised management of anal dysplasia. Lancet Oncol. 2013 Apr;14(4):273-4. doi: 10.1016/S1470-2045(13)70099-8. Epub 2013 Mar 15. No abstract available. PMID 23499545
- See also: Esser et al. DAIG-Leitlinie: Anale Dysplasien u. Analkarzinome bei HIV-Infizierten: Prävention, Diagnostik u. — http://www.awmf.org/uploads/tx_szleitlinien/055-007l_S1k_Anale_Dysplasien_Analkarzinom_HIV_infizierten_09-2013__01.pdf